CLINICAL TRIAL: NCT01724645
Title: Randomized, Open Label, Parallel Controlled, to Evaluate the Beneficial Effects of Korean Traditional Dites in Subjects With Hypertension and Type 2 Diabetes.
Brief Title: Beneficial Effects of Korean Traditional Diets in Subjects With Hypertension and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, director, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUH_KOREAN-FOOD_2-2_2010
Record Dates: First submitted 2012-10-29; First posted 2012-11-12 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Korean Traditional diets; hypertension; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Diabetes Mellitus | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Korean traditional diets (Experimental): Korean traditional diets (calorie 2,100kcal) for 12weeks
  Interventions: Dietary Supplement: Korean traditional diets
- Control group (Active Comparator): Control group : told to "eat as usal diet) for 12weeks
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Korean traditional diets — The consumption of Korean traditional diets reflecting the characteristics of Korean traditional diets without the limitation of calories has an effect on control of cardiovascular risk factor, so this study instructed all subjects of the intervention group to consume about 2,100kcal of served meals freely.
  The Korean Traditional diets, which encourages the intake of cooked rice, vegetables,soup,Kimchi and soy fermented foods.
  Other Names: The Korean Traditonal diets
  Arms: Korean traditional diets
Dietary Supplement: Control group — Told to " eat as usal diets".
  Other Names: Control diets
  Arms: Control group

SUMMARY:
This trial is being conducted to look for following changes when Korean traditional diets is taken in subjects with hypertension and type 2 diabetes:

To evaluate the improvement of the controlling fasting blood glucose and glycated hemoglobin.

To assess the controlling blood pressure and heart rate.

To evaluate the influence on cardiovascular risk factor, Triglyceride, cholesterol, High Density Lipoprotein-cholesterol and Low-Density Lipoprotein-cholesterol.

To evaluate the influence on Gamma-Glutamyl Transpeptidase.

To evaluate the influence on Cardiovascular risk factor.

To evaluate the influence on valsava score, breathing score and upright score.

DETAILED DESCRIPTION:
The investigators aimed to investigate the efficacy of Korean traditional diets in controlling fasting blood glucose fluctuation, blood pressure, and cardiovascular risk factors in hypertensive and type 2 diabetic patients who were taking medications prescribed for respective diseases in a 12-week.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are men and women volunteers 19~80years
* Subject who have hypertension and type 2diabetes.
* Subject who have taking oral medications :

(hypoglycemic, blood pressure and lipid modifying drugs).

* Subject must provide written informed consent to participate in the study.

Exclusion Criteria:

* Subject with a history or evidence of clinically significant gastrointestinal,anorectal, hepatic, renal, neurological, pulmonary, endocrine, blood tumor,psychiatric.
* Hypertension(DBP>116mmHg or SBP>200 mmHg) having the history of cardiovascular events or taking medications known to affect lipoprotein metabolism.
* Having Type 1 diabetes mellitus or uncontrolled Type 2 diabetes mellitus (HbA1c >9.0%).
* Subjects with the history of cancer.
* Subjects who have a gastrointestinal (GI) disease (Crohn's disease, etc.) that would increase the influence with absorbance medication or a GI surgery excluding appendectomy and hernia surgery.
* Having digestive, or central nervous system disorders.
* Subject is hematologic, or neuroretinopathy.
* Subject with uterine fibroids at ultrasonography.
* Having severe or malignant retinopathy.
* Having the impairment of renal and liver function, dysproteinemia, nephritic syndrome, or other renal disease.
* Having coagulopathy
* Having human immunodeficiency virus.
* Having the history of mental instability and of drug and alcohol.
* Having the history of reactions to our experimental products.
* Participating in other clinical trials within the past 2 months.
* Having laboratory tests, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study.
* Having the history of alcohol or substance abuse.
* Subject is pregnant, planning to become pregnant, or breast-feeding.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
HbA1C :Glycated Hemoglobin | 84days
  Glycated Hemoglobin is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.

SECONDARY OUTCOMES:
TG :Triglycerides | 84days
  Triglycerides is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
TC :Total cholesterol | 84days
  Total cholesterol is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
HDL-C :High Density Lipoprotein-Cholesterol | 84days
  HDL-C is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
LDL-C : Low Density Lipoprotein-Cholesterol | 84days
  LDL-C is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
Breathing score | 84days
  Breathing score is measured in study visits to the clinic, week 0(baseline)and week 12.
Valsalva score | 84days
  Valsalva score is measured in study visits to the clinic, week 0(baseline)and week 12.
Upright score | 84days
  Upright score is measured in study visits to the clinic, week 0(baseline) and week 12.
ApoA1 :Apolipoprotein A1 | 84days
  Apolipoprotein A1 is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
ApoB :Apolipoprotein B | 84days
  Apolipoprotein B is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
Apo E :Apolipoprotein E | 84days
  Apolipoprotein E is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
Free fatty acid | 84days
  Free fatty acid is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
Adiponectin | 84days
  Adiponectin is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
PAI-1 :Plasminogen activator inhibitor type 1 | 84days
  PAI-1 is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
Homocysteine | 84days
  Homocysteine is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
FPG :Fasting plasma glucose | 84days
  Fasting plasma glucose is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
DBP:Diastolic Blood Pressure | 84days
  DBP is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
SBP:Systolic Blood Pressure | 84days
  SBP is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
Heart rate | 84days
  Heart rate is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.

OTHER OUTCOMES:
weight | 84days
  weight is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
BMI:Body Mass Index | 84days
  BMI is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
Body fat percent | 84days
  Body fat percent is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
Waist | 84days
  Waist is measured in study visits to the clinic, week 0(baseline), week 4, week 8 and week 12.
Obesity associated gut microbiome(Bacteriodetes) | 84days
  Bacteriodetes is measured in study visits to the clinic, week 0(baseline)and week 12.
Obesity associated gut microbiome(Firmicutes) | 84days
  Firmicutes is measured in study visits to the clinic, week 0(baseline)and week 12.
Hypoglycemic(oral medication) | 84days
  Hypoglycemic oral medication is measured in study 0wk, 4wk, 8wk and 12wk.
Control blood pressure(oral medication) | 84days
  Control blood pressure(oral medication) is measured in study 0wk, 4wk, 8wk and 12wk.
Lipid modifying (oral medication) | 84days
  Lipid modifying (oral medication) is measured in study 0wk, 4wk, 8wk and 12wk.

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Wan Chae, MD., PhD, Study Director — Chonbuk National University Hospital
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea